CLINICAL TRIAL: NCT07251920
Title: Examination of the Dose-dependent Effects of Isometric Resistance Training on Decreases in Blood Pressure in Pre- and Hypertensive Adults
Brief Title: Isometric Resistance Training and Dose-dependent Effects in Pre- and Hypertensive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Northampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FREC2324002
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-01

CONDITIONS: Hypertension; Blood Pressure, High
Keywords: Hypertension; Blood pressure; Isometric contraction; Isometric resistance training; Isometric exercise
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Once-weekly training (Experimental): Performed isometric resistance training once per week (four 2-minute contractions).
  Interventions: Other: Isometric resistance training
- Twice-weekly training (Experimental): Performed isometric resistance training twice per week (eight 2-minute contractions).
  Interventions: Other: Isometric resistance training
- Thrice-weekly training (Active Comparator): Performed isometric resistance training thrice per week (12 2-minute contractions).
  Interventions: Other: Isometric resistance training

INTERVENTIONS:
Other: Isometric resistance training — isometric resistance training was performed on the chest, arms, and leg muscle groups using a band. Each contraction, was pulled at a perceived 30% (using a CR10 perceieved exertion rating scale) of maximum effort for 2 minutes; one repetition was performed using each muscle group. Weekly frequnecy changed between groups, ranging from once to thrice per week.

SUMMARY:
High blood pressure is prevalent in a third of the global population and is a key risk factor for cardiovascular disease, the leading cause of death. one lifestyle change that is recommended to reduce blood pressure is to exercise, typically by performing aerobic exercise, but this is often not well adhered to, given the physical and time demands associated with it. Isometric resistance training has been evidenced as an efficacious method to reduce blood pressure, even when performing four two-minute contractions per day, three days per week at 30% of maximum effort. At present, the dose-response effects have not been examined, which are required to identify the minimal effective dose, which could further reduce the temporal demands of this modality to potentially enhance adhernece even more in time-anxious individuals. Therefore, this study aimed to compare the efficacy of once- twice-, and thrice-weekly isometric resistance training programmes to lower blood pressure,

DETAILED DESCRIPTION:
The World Health Organisation have reported hypertension, a major risk factor for cardiovascular disease (CVD), strokes and coronary heart disease (CHD), to be near epidemic levels globally with over 30% of the world's population, at this time, suffering from hypertension. Over the past twenty years isometric resistance training (IRT) has been established as one of the best forms of nonpharmacological interventions for the prevention and treatment of hypertension and endorsed by the American College of Cardiology / American Heart Association in their most recent guidelines. Thrice weekly IRT programmes undertaken (4 x 2-minute isometric contractions) at 20-30% of an individual's maximum voluntary contraction (MVC) for a period of 4-10 weeks have demonstrated reductions in clinic resting and ambulatory systolic blood pressure (-4 to -10 mmHg), in both normotensive and hypertensive men and women with no reported difference in the magnitude of these reductions between women and men.

Whilst isometric training has been shown to produce clinically meaningful reductions in blood pressure, utilising the commonly used protocol (4 x 2-min contractions) three-times a week, one of the main barriers to therapeutic exercise interventions is time to undertake the intervention and despite the observed benefits, adherence and compliance tends to be low. Indeed, regular exercise adherence declines over time, with only 50% of individuals continuing with regular exercise within the first twelve months following the completion of a therapeutic treatment, with a lack of perceived time cited as one of the main barriers. With this in mind, it is important to determine the effects of training dose on the changes in blood pressure seen following IRT. To date there is very little research into the effects of IRT dose on resting blood pressure with only one study purposely investigated the area. Whilst to the authors knowledge no studies have investigated the effects of altered training dose on ambulatory or diurnal blood pressure variations. Although three times a week has become the most commonly applied protocol there is no evidence to confirm that it is the most efficacious. As training dose is an important determinant of adaptations to exercise training, and with a lack of time cited as a perceived barrier to undertaking exercise, there is a need to determine the most efficacious training protocol to elicit clinical reductions in blood pressure, including shorter time saving (once or twice weekly) protocols.

Therefore, the study aims are to determine if a reduction in the weekly dose of isometric training, such as a reduction in the number of total contractions and therefore a reduced time commitment (once or twice weekly) would produce a similar hypotensive response to those reported.

ELIGIBILITY:
Inclusion Criteria:

* not taking anti-hypertensive medication
* borderlerine hypertensive or hypertensive (systolic blood pressure >139 mmHG, diastolic blood pressure > 89 mmHg

Exclusion Criteria:

* conditoned to resistance training
* currently taking anti-hypertensive medication
* regularly smoke or vape
* are pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure | Through study completion (12 weeks)
  Blood pressure assessed during a 24-hour window

SECONDARY OUTCOMES:
Resting blood pressure | Through study completion (12 weeks)
  Blood pressure taken following a 10-minute rest period

CONTACTS AND LOCATIONS:
Locations (1):
- University of Northampton, Waterside Campus, Northampton, Northamptonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be uplaoded to a reposiotory hosted by The University of Northampton and will be publicly available online. The DOI and URL to the data set will be included in future publications.
Supporting Information: Study Protocol
Time Frame: IPD will be available when the study is published.
Access Criteria: Data underlying the findings of the study will be publicly available via a repository.

REFERENCES:
- [Background] Smart NA, Way D, Carlson D, Millar P, McGowan C, Swaine I, Baross A, Howden R, Ritti-Dias R, Wiles J, Cornelissen V, Gordon B, Taylor R, Bleile B. Effects of isometric resistance training on resting blood pressure: individual participant data meta-analysis. J Hypertens. 2019 Oct;37(10):1927-1938. doi: 10.1097/HJH.0000000000002105. PMID 30889048
- [Background] Lopes S, Felix G, Mesquita-Bastos J, Figueiredo D, Oliveira J, Ribeiro F. Determinants of exercise adherence and maintenance among patients with hypertension: a narrative review. Rev Cardiovasc Med. 2021 Dec 22;22(4):1271-1278. doi: 10.31083/j.rcm2204134. PMID 34957769
- [Background] Zhou B, Perel P, Mensah GA, Ezzati M. Global epidemiology, health burden and effective interventions for elevated blood pressure and hypertension. Nat Rev Cardiol. 2021 Nov;18(11):785-802. doi: 10.1038/s41569-021-00559-8. Epub 2021 May 28. PMID 34050340
- [Background] Garcia-Hermoso A, Lopez-Gil JF, Ramirez-Velez R, Alonso-Martinez AM, Izquierdo M, Ezzatvar Y. Adherence to aerobic and muscle-strengthening activities guidelines: a systematic review and meta-analysis of 3.3 million participants across 32 countries. Br J Sports Med. 2023 Feb;57(4):225-229. doi: 10.1136/bjsports-2022-106189. Epub 2022 Nov 23. PMID 36418149